CLINICAL TRIAL: NCT05058781
Title: Evaluation of Minipuberty in Infants Born With a Variation in Sexual Development
Brief Title: Minipuberty in Infants Born With Potential Hypogonadism Hypogonadotrope
Acronym: MiniNO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Nelly Pitteloud, Professor, Head od Endocrine department, Centre Hospitalier Universitaire Vaudois
Other Study IDs: CER-VD 2016-01232
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: DSD; CHH

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Biospecimen Retention: Samples With DNA — blood, urine, buccal swabs, cord blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Disorders of sex development (DSD) occur in 1/3000 births and are defined by variation in aspect of external genital organs, e.g. cryptorchidism, hypospadias and micropenis in male infants and clitoral hypertrophy in female infants. Genetic, hormonal and environmental factors are implicated in DSD. Infants with congenital hypogonadism hypogonadotrope (CHH) can present with DSD. Evaluation of hormonal profile during minipuberty could be of great help to better characterize the etiology of DSD and CHH in particular. Our main objective is to study hormonal profile during the minipuberty of infants born with DSD or born from parents with CHH compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* infants born with symptoms of DSD
* infants born from parents with CHH

Exclusion Criteria:

* premature < 35 weeks of gestation
* male infants with high scrotal cryptorchidism

Max Age: 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All infants born in canton de Vaud in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Hormonal changes in blood and in urine during minipuberty (LH, FSH, steroid profile, Testosterone, Estradiol (in girls), AMH, inhibin B) | at 2, 6 and 9 months of age (window for minipuberty)
  Reproductive profile:
  LH and FSH (UI/L) steroid profile (nmol/L) Testosterone and Estradiol (nmol/L) AMH (ng/mL) inhibin B (pg/mL)

SECONDARY OUTCOMES:
quantification of Nitric Oxide metabolites during minipuberty | at 2, 6 and 9 months of age
  measurements of Nitrite (NO2-) and nitrate (NO3-) in blood
change in expression of genes involved in the NO pathway | at birth (if available), 2, 6 and 9 months of age
  RNA sequencing of samples collected in blood

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Pitteloud, MD, Principal Investigator — CHUV
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland